CLINICAL TRIAL: NCT01165008
Title: Anakinra in Patients With Refractory Idiopathic Inflammatory Myopathies
Brief Title: Anakinra in Myositis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Ingrid Lundberg, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: KS 01; 03-144 (Other: Etikprovningsnamnden i Stockholm)
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2010-07-19 (Estimated); Status verified 2005-02

CONDITIONS: Polymyositis; Dermatomyositis; Inclusion Body Myositis
MeSH Terms: conditions — Polymyositis; Dermatomyositis; Myositis, Inclusion Body | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Anakinra

SUMMARY:
To investigate the effect of the interleukin-1 (IL-1) blocking agent, anakinra, in patients with treatment-resistant inflammatory myopathies.

Patients and methods: Fifteen patients with refractory polymyositis (PM), dermatomyositis (DM), or inclusion body myositis (IBM) were treated with 100 mg anakinra subcutaneously per day during 12 months. Outcome measures included myositis disease activity score with improvement defined according to The International Myositis Assessment and Clinical Studies Group (IMACS) and for muscle performance the functional index of myositis (FI). In addition repeat muscle biopsies were performed

ELIGIBILITY:
Inclusion Criteria:

Men and women aged 18 to 80 years with diagnosis of PM, DM or IBM based Peter and Bohan's and Grigg's criteria. All patients had to be capable of giving informed consent. Other inclusion criteria were muscle strength and/or function reduced at least 20 % below predicted values as measured by functional index (FI) [45-47] and failure to respond to treatment with high-dose glucocorticoids (0.75 mg/kg/day for at least one month) in combination with azathioprine and/or methotrexate for at least two months.

-

Exclusion Criteria:

serious infections such as hepatitis, pneumonia, pyelonephritis in the previous 3 months; history of opportunistic infections such as tuberculosis, drug resistant atypical mycobacterium, active pneumocystis carinii, active cytomegalovirus infection; documented HIV infection; alcoholism, alcoholic liver disease or other chronic liver disease; chest x-ray suggestive of active tuberculosis; and pregnant, nursing mothers or patients with planned pregnancy within one and a half years of enrolment.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-09; Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden